CLINICAL TRIAL: NCT05112874
Title: ImmuneSense™ COVID-19 Cross-Reactivity Study
Status: Withdrawn | Type: Observational
Why Stopped: Flu season over.
Sponsor: Adaptive Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-00822
Record Dates: First submitted 2021-10-27; First posted 2021-11-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Coronavirus Disease; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Seasonal Coronavirus; Upper Respiratory Tract Infection
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cross-Reactive Cohort: Ages 18-89, Exhibiting symptoms compatible with a viral upper respiratory tract infection at the time of screening.
  Lab test confirming
  1. Negative for SARS-CoV-2 (by Polymerase Chain Reaction (PCR) or Antibody detection test)
  2. Respiratory Panel positive for the common seasonal coronaviruses: NL63, 229E, OC43, and HKU1

SUMMARY:
Adaptive Biotechnologies has developed a clinical test called T-Detect COVID Test that can identify a T-cell response to the SARS-CoV-2 virus, indicating recent or prior infection This study aims to evaluate the potential cross-reactivity of the T-Detect COVID test in participants presenting with viral upper respiratory tract infections within the assay's intended use population and testing positive for seasonal coronavirus.

DETAILED DESCRIPTION:
Prospective ascertainment of a minimum of 10 individuals exhibiting symptoms of viral upper respiratory tract infections, between the ages of 18-89 residing within the United States and being tested for SARS-CoV-2 infection during the 2021-2022 cold and flu season (~Nov. 2021 - May 2022).

Participants will complete an electronic screening questionnaire to determine eligibility, be consented, and scheduled for a study visit that will be conducted by study staff or mobile phlebotomist. The identification and recruitment of participants will protect privacy and be free of undue influence. Biological samples, including blood samples and nasopharyngeal swabs, will be collected via mobile phlebotomy in participant's homes with proper safety precautions in place. Study metadata and questionnaire information will be self-reported and/or recorded by study staff as applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Exhibiting viral upper respiratory infection symptoms during the symptomatic phase of infection and tested positive for a common seasonal coronavirus (NL63, 229E, OC43, and HKU1) at time of diagnosis for initial symptoms
2. Available for specimen collection greater than 14 days and less than 100 days after first exhibiting symptoms of confirmed seasonal coronavirus infection.
3. Male and female participants of any race and ethnicity between 18 to 89 years of age (inclusive) at the time of enrollment in the study
4. Able to communicate with the investigator, understand, and comply with the requirements of the study

Exclusion criteria:

1. Did not develop symptoms related to their diagnosed seasonal coronavirus infection
2. Prior diagnosis of COVID-19 or any positive test result for SARS-CoV-2 infection or antibodies test
3. Cohabitated with or has had significant exposure (per the Center for Disease Control guidelines) to another individual with known COVID-19
4. Protected populations including pregnant women, prisoners, mentally disabled persons, and wards-of-the state.
5. Any significant condition, laboratory abnormality, or psychiatric illness that would prevent the participant from safely participating in the study
6. Donated more than 500cc or 1 pint of blood in the past 60 days prior to the study blood draw
7. Received a COVID-19 vaccine, including a single dose of a multiple dose vaccine regimen
8. Participated in a COVID-19/SARS-CoV-2 study or received a SARS-CoV-2 antibody, or other SARS-CoV-2 therapeutic investigational drug or compound that will impact results of the study at the discretion of the investigator, such as but not limited to a SARS-CoV-2 antibody, therapeutic, or other medication that may impact the person's immune response

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruiting individuals ages 18-89 at the time of screening are exhibiting symptoms compatible with a viral upper respiratory tract infection and obtain negative test result for SARS-CoV-2. Eligible participants must also test positive for one of the following common seasonal coronaviruses: NL63, 229E, OC43, and HKU1 via Respiratory Panel test.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Cross-Reactivity of T-Detect COVID | 15-100 days from symptoms onset
  Adaptive Biotechnologies Corporation has developed a clinical test called T-Detect COVID, which is intended to identify a T-cell response to the SARS-CoV-2 virus, indicating recent or prior infection.
  This study will assess the clinical performance of the T-Detect COVID test in participants presenting with symptoms of a viral upper respiratory tract infections.
  Eligible participants must have proof of negative result from an Emergency Use Authorization approved Reverse transcription-polymerase chain reaction (RT-PCR) assay and positive result with Clinical Laboratory Improvement Amendment (CLIA) validated assay for other seasonal coronaviruses.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Gill, Principal Investigator — Adaptive Biotechnologies
Locations (1):
- Adaptive Biotechnologies, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No